CLINICAL TRIAL: NCT02522169
Title: Verbessertes Therapiemanagement für pädiatrische CED-Patienten Mit Chronisch-entzündlicher Darmerkrankung: Eine Randomisierte Multizentrische Studie, Welche Die Effektivität Einer Talspiegel-gesteuerten Infliximab-Erhaltungsphase Mit Dem herkömmlichen Dosierungsregime Vergleicht Trough Level Optimized Pediatric Inflammatory Bowel Disease Therapy: A Randomized Multicenter Study Comparing Effectiveness of Trough Level Optimized Infliximab Maintenance Therapy With Standard Dosing Regimen of Pediatric Patients With Crohn's Disease
Brief Title: TOPIT; Trough Level Optimized Pediatric Inflammatory Bowel Disease Therapy: A Multicenter Study Comparing Effectiveness of Trough Level Optimized Infliximab Maintenance Therapy With Standard Dosing Regimen of Pediatric Patients With Crohn's Disease
Acronym: TOPIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Klinikum Westbrandenburg GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-000076-25
Record Dates: First submitted 2015-05-03; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Pediatric Crohns Disease
MeSH Terms: interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional treatment (Active Comparator): The patients of the control group undergo Infliximab-maintenance according to the approved dosing scheme, initially with 5 mg/kg body weight Infliximab. Before each administration laboratory parameters will be controlled (Albumin, CrP, Calprotectin) and disease activity scores will be obtained (PCDAI / PUCAI). Infliximab trough levels will be assessed but not have any implication. In the presence of clinical signs of a disease exacerbation and after exclusion of other causes an adjustment of the dosage will follow for the next Infliximab-infusion:
  A) interval shortening, or B) Dose increase to 10 mg / kg body weight. With a clinical stable course of the disease without signs of deterioration, the dosage and the eight-week interval will be maintained.
  Interventions: Drug: Infliximab
- Intervention Group (Experimental): Aiming to maintain the therapeutic window of Infliximab a de- or increase of the dose or infusion interval will be carried out for the following administration, provided the patient shows no signs of a clinical worsening. With good trough levels and clinically stable conditions the therapy will be continued without modification until next check-up. In the case of an eminent disease exacerbation Infliximab trough levels and the search for anti - Infliximab antibodies should guide further treatment decisions. With trough levels below the target range antibody testing should be performed.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — This is a randomized, prospective, parallel -controlled study, simple blinded and multicenter designed. Study centers are the Department of Child and Adolescent Medicine of the Ernst von Bergmann Hospital, Potsdam, and the Department of Child and Adolescent Medicine of Charité, Berlin.
  We estimate a sample size of 50 patients per center. Study inclusion begins with given consent of the patient and the legal guardian. Patients will be randomized in control- and intervention group separately for Cohn's disease. An equal age and gender distribution is targeted for both control and intervention group. Sub groups will be formed depending on the time span from completed Infliximab induction to study enrollment (group A< 6month, group B < 6 month). Observation period is one year.
  Other Names: Remicade

SUMMARY:
This clinical trail intends to evaluate interventions based on the Infliximab trough levels for an individualized therapy adaption for pediatric IBD-patients undergoing anti-TNF-alpha-therapy. Main aim of the individualized strategy is to attain and maintain early disease control in order to keep as many patients as possible in disease remission, and to avoid primary and secondary therapy failure.

DETAILED DESCRIPTION:
Anti TNF-alpha agents such as Infliximab are efficient and safe in treating pediatric IBD-patients. However maintaining the remission and therapeutic response is still a challenge for the practitioner. In addition to a relevant number of primary non-responding patients individual clearance and immunogenic effects lead to secondary loss of response in a significant number of patients. So far these patients are clinically managed by decrease of the infusion interval or increasing the dose. Besides an increased risk for potential side effect a high number of patients need to switch treatment to other biologicals despite interventions. Improved strategies are needed to avoid primary and secondary therapeutic failure, and a promising lead seems to be the individualized therapy.

Especially in pediatric IDB-patients with faster turnover of anti-TNF based on a higher metabolism rate new ways of adapting the dose and maintaining therapeutic serum levels are necessary. In this context the role of IFX-trough levels is not fully clear. Previous studies have shown that serum IFX trough levels correlate inversely with the turnover rate and directly to therapeutic response. Thus it is highly desirable to keep trough levels in therapeutic window. In adult patients recent studies have shown advantages in using IFX-trough levels for therapy optimization, leading to better disease control in short and long term. However there is until now no clear evidence that shows benefits for an IFX-target-level approach during the maintenance of therapy.

An early therapy optimization from the beginning on with rapid control of mucosal inflammation seems to set the pathway for sustained therapy response and disease remission.

We assume a clear benefit for an individualized, IFX-trough-level guided therapy optimization for pediatric IDB-patients and intend to clarify the role of Infliximab trough levels in this planned trial.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients of both sexes with Cohn's disease
* Assured diagnosis of Cohn's disease according to the Porto criteria
* Regular attendance of gastroenteric consultations at one of the study centers
* Minimum patients age of 6 years, maximum age of 16 years
* Infliximab therapy with permitted / without co- medication
* Completed induction with Infliximab in accordance to the approved conventional scheme with primary therapy response
* Written consent of the patient and the legal guardian

Exclusion Criteria:

* No consent of the patient and / or legal guardian
* Serious side effects under Infliximab therapy in the past
* Primary non-responder to Infliximab after first three cycles

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
disease remission | 12 months
  The trial's primary endpoint is the disease remission of pediatric patients receiving Infliximab therapy after an observation period of twelve month. This will be done by comapring the PCDAI of both groups after 12 month and the PCDAI perfomance in the respective group during the observation period.
  For monitoring the disease activity the PCDAI (Pediatric Crohn's Disease Activity Index) is deployed.

SECONDARY OUTCOMES:
Secondary endpoint is the rate of adverse reactions | 12 months
  safety
Costs of treatment | 12 months
The number of patients with a reset of therapy due to secondary loss of response, e.g. to a differend biological therapy, is the focus of ths secondary outcome | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Augustin Gonçalves, Principal Investigator — Klinikum Westbrandenburg